CLINICAL TRIAL: NCT03171935
Title: Wean Early With High-Flow Nasal Cannula Oxygenation Versus Noninvasive Positive Pressure Ventilation in Patients With Acute Hypoxemic Respiratory Failure: a Multicenter, Randomized, Controlled Trial (the WHEN Study)
Brief Title: Wean Early With HFNCO vs NPPV in Patients With AHRF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Zujin Luo, MD, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BeijingCYH-ICU-005
Record Dates: First submitted 2017-05-29; First posted 2017-05-31 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Patients With Acute Hypoxemic Respiratory Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-Flow Nasal Cannula Oxygenation (Experimental)
  Interventions: Device: High-Flow Nasal Cannula Oxygenation
- Noninvasive Positive Pressure Ventilation (Experimental)
  Interventions: Device: Noninvasive Positive Pressure Ventilation
- Conventional Weaning (Active Comparator)
  Interventions: Device: Conventional weaning

INTERVENTIONS:
Device: High-Flow Nasal Cannula Oxygenation — High-flow nasal cannula oxygenation will be applied immediately after early extubation, with a gas flow rate of 50 liters per minute and a fraction of inspired oxygen of 1.0 at initiation. The fraction of inspired oxygen will be subsequently adjusted to maintain a peripheral oxygen saturation of 92% or more.
  Arms: High-Flow Nasal Cannula Oxygenation
Device: Noninvasive Positive Pressure Ventilation — Noninvasive positive pressure ventilation will be applied immediately after early extubation, with a noninvasive ventilator (Respironics V60, Philips) using the NIPSV mode at initiation. The fraction of inspired oxygen will be adjusted to achieve SpO2 >92% with an initial expiratory positive airway pressure (EPAP) of 4 cmH2O. EPAP will be increased gradually in increments of 1-2 cmH2O, up to a maximum of 12 cmH2O, to achieve SpO2 >96%. Inspiratory positive airway pressure (IPAP) will be initially set at 8 cmH2O and be increased gradually in increments of 1-2 cmH2O according to patients' tolerance to obtain a tidal volume (VT) of 6-8 mL/kg.
  Arms: Noninvasive Positive Pressure Ventilation
Device: Conventional weaning — The patients will undergo conventional weaning protocol. Extubation and subsequent oxygen therapy with venturi mask will be performed after successful spontaneous trial.
  Arms: Conventional Weaning

SUMMARY:
The main purpose of the present study is to verify whether, as compared with conventional weaning, early weaning with high-flow nasal cannula oxygenation or noninvasive positive pressure ventilation may more effective in shortening the duration of invasive ventilation, hence reducing the rates of complications and mortality in patients with acute hypoxemic respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

1. Orotracheal intubation；
2. PaO2 <60mmHg（venturi mask，FiO2=0.5），and PaCO2 ≤45mmHg；
3. Meeting criteria for weaning readiness；
4. Spontaneous breathing trial failure.

Exclusion Criteria:

1. Age<18；
2. Duration of invasive ventilation <48h；
3. Tracheotomy；
4. Percentage of cuff leak volume in tidal volume<15.5%；
5. Unable to spontaneously clear secretions from their airway；
6. Recent oral，nasal，facial or cranial trauma or surgery；
7. Recent gastric or esophageal surgery；
8. Active upper gastro-intestinal bleeding；
9. Severe abdominal distension；
10. Lack of co-operation；
11. Chronic respiratory disease such as chronic obstructive pulmonary disease, asthma, interstitial lung disease and neuromuscular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Duration of invasive mechanical ventilation | 2.5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Institute of Respiratory Medicine, Department of respiratory and critical care medicine, Beijing Chao-Yang Hospital Jingxi Campus, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No